CLINICAL TRIAL: NCT02954315
Title: The Effect of Almonds on Skin Lipids and Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 930524
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Almond arm (Experimental): The almond dose will be provided as 20% of total energy (20% E) in the diet. This dose was selected based on a previous randomized trial examining lipid parameters in response to 0, 10%, and 20% E as dietary almonds and a recent meta-analysis of intervention trials.
  Interventions: Other: Almonds
- Western diet Snack (Granola bar + Pretzels) (No Intervention): The control snack will be a typical western diet snack (see Table 1). The calorie-matched control snack will be commercially available individually wrapped food products such as a small granola bar + pretzels.

INTERVENTIONS:
Other: Almonds
  Arms: Almond arm

SUMMARY:
Investigators hypothesize that regular consumption of almonds will augment the long chain fatty acid profile and the alpha-tocopherol levels, improve the skin barrier function, and improve the appearance of facial wrinkles in post-menopausal women.

DETAILED DESCRIPTION:
Primary Endpoint:

A) Change in wrinkle depth. Full facial photographs will be obtained at baseline, 8 weeks, and 16 weeks. The images will be obtained with the 3D Clarity Pro® Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA) that has standardized positioning and lighting. This system can assess average wrinkle depth. The PI has already validated this measurement tool against standard clinical grading of facial wrinkles[13].

Secondary Endpoint:

A) Change in clinical appearance of facial wrinkles on lateral canthi: Two blinded dermatologists will grade the photographs obtained at each of the time points on the lateral canthi ("crow's feet"). The dermatologists will not know which group the subjects were in.

B) Change in facial sebum production through the use of a Sebumeter, a commonly used device that measures sebum excretion rate [13,17]. Sebum excretion rate will be measured at baseline, 8 weeks, and 16 weeks.

C) Change in serum and sebum lipid profiles obtained through the use of Sebutapes at baseline, 8 weeks, and 16 weeks.

D) Change in the serum and sebum lipid profile for assessment of long chain/short chain fatty acid ratios and the NS ceramide content.

Procedures Involved This study will be a 16-week supplementation study that utilizes two study groups: 1) Control group 2) Almond supplementation: 20% energy intake. This will be a randomized, rater-blinded, controlled study.

There will be a total of 30 subjects:

Control Group: n=15 Almond Supplementation: n=15

The subjects will be recruited from the UC Davis Dermatology Department, the surrounding clinics in a 25 mile radius, and the general population in the Davis and Sacramento areas. The greater Sacramento area has a population of over 2 million to draw from and recruitment will be conducted through the use of Social Media and flyer based recruitment.

Investigators will collect medical history and current medications from study participants- this is outlined in the HIPAA form. The two intervention groups will consist of those receiving almonds and those that are receiving a calorie matched snack. The almond dose will be provided as 20% of total energy (20% E) in the diet. This dose was selected based on a previous randomized trial examining lipid parameters in response to 0, 10%, and 20% E as dietary almonds and a recent meta-analysis of intervention trials of tree nuts [23,24]. The control snack will be a typical western diet snack. The calorie-matched control snack will be commercially available individually wrapped food products such as a small granola bar + pretzels. Once a subject has met inclusion criteria and has signed IRB consent, anthropometric data will be obtained, 3-24 hour recall will be collected by phone, skype, or in person by a Registered Dietitian, training will be provided for recording dietary records, and estimated caloric needs will be calculated. Estimated energy needs (EER) will be determined using the Mifflin-St. Jeor equation and total daily energy needs (TDE) calculated as EER x activity factor of 1.3-1.5 for sedentary to average activity, or a higher activity level as indicated. A representative example of a 60 year old woman, 5'4", 140 pounds with typical activity level yields TDE of approximately 1,600 - 1,800 kcal/day, and 20% E of 320-360 kcal/day. The dose of almonds would be 2 ounces (equal to 23 whole kernels)/day, providing 328 calories.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Fitzpatrick skin types 1 and 2
* Able to follow dietary intervention and attend all study visits

Exclusion Criteria:

* Those with a nut allergy
* Smoking:

  * Current smokers
  * Those that have smoked within the past year
  * Former smokers with greater than a 20 pack-year history of smoking within the past 20 years will be excluded.
* Those with an autoimmune photosensitive condition or a known genetic condition with a deficiency in collagen production (such as Ehler-Danlos)
* Those that already obtain 20% of their energy intake from nut consumption
* Those with implausible reported energy intakes of <1,000 kcal/d or >3,000 kcal/d
* Individuals who are unwilling to discontinue high antioxidant supplements and daily food sources listed below, during the washout and intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in wrinkle depth | 16 weeks

SECONDARY OUTCOMES:
Change in clinical appearance of facial wrinkles on lateral canthi | 16 weeks
Change in facial sebum production through the use of a Sebumeter | 16 weeks
Change in serum and sebum lipid profiles | 16 weeks
Change in the serum and sebum lipid profile for assessment of long chain/short chain fatty acid ratios and the NS ceramide content | 16-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, M.D., Principal Investigator — UC Davis
Locations (1):
- UC Davis Department of Dermatology, Clinical Trials Unit, Sacramento, California, United States

REFERENCES:
- [Background] Alasalvar C, Bolling BW. Review of nut phytochemicals, fat-soluble bioactives, antioxidant components and health effects. Br J Nutr. 2015 Apr;113 Suppl 2:S68-78. doi: 10.1017/S0007114514003729. PMID 26148924